CLINICAL TRIAL: NCT01306721
Title: A Randomized, Double Blind, Parallel Group Study for Assessing the Efficacy and Safety of a Twice-daily Fexofenadine HCl 60 mg - Pseudoephedrine HCl 60 mg Combination or Fexofenadine HCl 60 mg - Pseudoephedrine HCl 120 mg Combination Versus Allegra® 60 mg in Patients With Seasonal Allergic Rhinitis
Brief Title: Fexofenadine HCL - Pseudoephedrine HCL Combination Versus Allegra in Patients With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC11243; U1111-1115-7613 (Other: UTN)
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Rhinitis Seasonal
MeSH Terms: interventions — fexofenadine; Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- FEX 60 mg (Active Comparator): Study medications is administered one hour before or two hours after a meal twice a day.
  Placebo lead-in period: 1 placebo tablet of fexofenadine 60 mg + 2 placebo tablets of fexofenadine 60 mg/pseudoephedrine 60 mg (fixe dose combination)
  Double-blind treatment period:
  1 tablet of fexofenadine 60 mg + 2 placebo tablets of fexofenadine 60 mg /pseudoephedrine 60 mg (fixe dose combination)
  Interventions: Drug: fexofenadine HCL (M016455); Drug: pseudoephedrine; Drug: fexofenadine HCL matching placebo; Drug: pseudoephedrine matching placebo
- FEX 60 mg/PSE 60 mg (Experimental): Study medications is administered one hour before or two hours after a meal twice a day.
  Placebo lead-in period: 1 placebo tablet of fexofenadine 60 mg + 2 placebo tablets of fexofenadine 60 mg/pseudoephedrine 60 mg (fixe dose combination
  Double-blind treatment period:
  1 tablet of fexofenadine 60 mg/pseudoephedrine 60 mg (fixe dose combination) + 1 placebo tablet of fexofenadine 60 mg / pseudoephedrine 60 mg (fixe dose combination)
  Interventions: Drug: fexofenadine HCL (M016455); Drug: pseudoephedrine; Drug: fexofenadine HCL matching placebo; Drug: pseudoephedrine matching placebo
- FEX 60 mg/PSE 120 mg (Experimental): Study medications is administered one hour before or two hours after a meal twice a day.
  Placebo lead-in period: 1 placebo tablet of fexofenadine 60 mg + 2 placebo tablets of fexofenadine 60 mg/pseudoephedrine 60 mg (fixe dose combination)
  Double-blind treatment period:
  2 tablets of fexofenadine 30 mg/pseudoephedrine 60 mg (fixe dose combination) + 1 placebo tablet of fexofenadine 30 mg
  Interventions: Drug: fexofenadine HCL (M016455); Drug: pseudoephedrine; Drug: fexofenadine HCL matching placebo

INTERVENTIONS:
Drug: fexofenadine HCL (M016455) — Pharmaceutical form:tablet Route of administration: oral
Drug: pseudoephedrine — Pharmaceutical form:tablet
  Route of administration: oral
Drug: fexofenadine HCL matching placebo — Pharmaceutical form:tablet
  Route of administration: oral
Drug: pseudoephedrine matching placebo — Pharmaceutical form:tablet
  Route of administration: oral
  Arms: FEX 60 mg; FEX 60 mg/PSE 60 mg

SUMMARY:
Primary Objective:

- To evaluate the efficacy on the nasal congestion of a twice-daily fexofenadine HCl 60 mg - pseudoephedrine HCl 60 mg combination (FEX60/PSE60) and fexofenadine HCl 60 mg - pseudoephedrine HCl 120 mg combination (FEX60/PSE120) versus fexofenadine HCl 60 mg (FEX60) in patients with seasonal allergic rhinitis (SAR).

Secondary Objectives:

* To evaluate the efficacy of a twice-daily FEX60/PSE60 and FEX60/PSE120 versus FEX60 on nasal symptoms (sneezing, rhinorrhea, and nasal congestion), eye symptom, and daily activity impairment.
* To assess the safety of a twice-daily FEX60/PSE60 and FEX60/PSE120 versus FEX60.

DETAILED DESCRIPTION:
The study duration for each patient is 3 weeks and 3 days:

1. Lead-in period: 1 week
2. Treatment period: 2 weeks
3. Follow-up period: 3 days

ELIGIBILITY:
Inclusion criteria:

- Patients with seasonal allergic rhinitis (SAR): Patients with a history of SAR symptoms during the season when cedar pollen levels are increased for at least 2-years

Exclusion criteria:

* At the start of the placebo lead-in period:

  * Patients who are negative for IgE Antibody test
  * Expected nasal congestion score is less than 2
* The last 3 days of the lead-in period:

  * Nasal congestion scores are 2 or more and not all 4
  * Patients with all nasal symptoms (sneezing, rhinorrhea, and nasal congestion). A total score for nasal symptoms (sneezing, rhinorrhea, and nasal congestion) and eye symptom is less than 6
  * Patients with 2 or more nasal symptoms (sneezing and rhinorrhea) and eye symptoms score is 4

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Changes in the nasal congestion score based on the patient's symptom diary | over 2 treatment weeks (from baseline to end of treatment)

SECONDARY OUTCOMES:
Changes in the total score of 4 symptoms, each nasal symptom (sneezing, rhinorrhea, and nasal congestion) and eye symptom | over 2 treatment weeks (from baseline to end of treatment)
Changes in total score of 4 symptoms on a daily, day-time, and night-time bases | over 2 treatment weeks (from baseline to end of treatment)
Changes in each symptom (sneezing, rhinorrhea, nasal congestion, and eye symptoms) score and the daily activity impairment score | over 2 treatment weeks (from baseline to end of treatment)
Changes in each symptom score and the daily activity impairment score on a daily, day-time and night-time basis | over 2 treatment weeks (from baseline to end of treatment)
Nasal findings | over 2 treatment weeks (from baseline to end of treatment)
Patient's impression | over 2 treatment weeks (from baseline to end of treatment)
Patient's safety | over 2 treatment weeks (from baseline to end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Japan (3):
  - Investigational Site Number 392002, Koganeishi
  - Investigational Site Number 392003, Osaka
  - Investigational Site Number 392001, Shinjuku-Ku